CLINICAL TRIAL: NCT05402605
Title: The Effectiveness and Safety of Artificial Oocyte Activation With Calcium Ionophore in Low Prognosis Women Classified as POSEIDON Group 4: a Randomized Clinical Trial
Brief Title: AOA Versus Non-AOA in Low Prognosis Patients by the POSEIDON Criteria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/2022/MĐ-HĐĐĐ
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: in Vitro Fertilization
Keywords: POSEIDON; in vitro fertilization; live birth; low prognosis; AOA
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI with AOA (Active Comparator): The oocytes were transferred into the calcium ionophore activation solution for two times of post-ICSI AOA (Ionomycin concentration of 10 µM).
  Then the oocytes will be washed several times using the medium drops in dish AOA and dish ICSI, then divided into drops with maximum 3 oocytes per drop for culturing. After that, the culture dish will be put in the K-system G185 incubator at 37oC, 6% CO2, and 5% O2.
  Interventions: Procedure: ICSI with AOA
- ICSI without AOA (Active Comparator): Post-ICSI oocytes will be cultured in drops containing the Sage - 1 - StepSM medium (maximum 3 oocytes per drop) at 37oC, 6% CO2 and 5% O2 in K-system G185 incubator.
  Interventions: Procedure: ICSI without AOA

INTERVENTIONS:
Procedure: ICSI with AOA — Step 1: All post-ICSI oocytes will be added in the medium drop in AOA dish, these oocytes will be placed in the incubator at 37oC, 6% CO2, and 5% O2 for 20 minutes.
  Step 2: After 20 minutes, calcium ionophore stock (Sigma-Aldrich - USA) will be diluted into 10µM drops in AOA dish.
  Step 3: After 10 minutes of incubation, all post-ICSI oocytes will be moved to the AOA drop, then this dish will be put back in the incubator for 10 minutes.
  Step 4: After 10 minutes, all the oocytes in drop AOA will be moved to another drop for rinsing and then put back in the incubator for 20 minutes.
  Step 5: After 20 minutes, the oocytes will be moved into drop AOA and then put back in the incubator for 10 minutes.
  Step 6: After 10 minutes, all post-ICSI oocytes will be added in the medium drop, then divided into drops with maximum 3 oocytes per drop for culturing. After that, the culture dish will be put in the K-system G185 incubator at 37oC, 6% CO2, and 5% O2
  Arms: ICSI with AOA
Procedure: ICSI without AOA — Conventional ICSI procedure will be performed without the application of AOA.
  Arms: ICSI without AOA

SUMMARY:
Poor ovarian response (POR) remains one of the significant challenges of Assisted Reproductive Technology (ART). Facing difficulties related to clinical practice, optimizing the embryo culture process is necessary to improve the embryo number and quality in this group of patients. Potential techniques mentioned in the current literature include follicular size at trigger, dual trigger, artificial oocyte activation (AOA), blastocyst transfer, and the role of preimplantation genetic testing for aneuploidy (PGT-A). AOA is currently expected to improve treatment outcomes in poor ovarian responders with the potential for clinical efficacy. However, this issue has not been evaluated before.

DETAILED DESCRIPTION:
Poor ovarian response (POR) remains one of the significant challenges of Assisted Reproductive Technology (ART). Patients with POR yield a low number of oocytes, leading to a low number of useable embryos and a decline in the live birth rate. According to the consensus of the European Society of Human Reproduction and Embryology (ESHRE) in 2011, POR was diagnosed using Bologna criteria. However, some recent studies show the classification by Bologna is not efficient, because the oocyte number should be combined with female age since the likelihood of achieving a live birth among patients with similar oocyte yield ultimately depends on the age of the patient. In 2016, POSEIDON (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number) Group was established and released the new criteria. The POSEIDON criteria proposed a shift from the terminology of POR to the concept of low prognosis. According to POSEIDON criteria, low prognosis account for 30-40% of all stimulated in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) cycles. The low prognosis patient is classified into four groups according to the results of ovarian reserve markers (AMH, AFC, or both), female age, and the number of oocytes retrieved in previous cycles, such as: maternal age < 35, AMH ≥ 1,2 ng/ml and AFC ≥ 5 (subgroup 1a: < 4 oocytes; subgroup 1b: 4-9 oocytes); maternal age ≥ 35, AMH ≥ 1,2 ng/ml and AFC ≥ 5 (subgroup 2a: < 4 oocytes; subgroup 2b: 4-9 oocytes); maternal age < 35, AMH < 1,2 ng/ml and AFC < 5; maternal age ≥ 35, AMH < 1,2 ng/mL and AFC < 5. Although many efforts have been made to improve treatment outcomes in this group of patients, such as researching, understanding, and modifying clinical ovarian stimulation regimens, the results are still not feasible. Especially, group 4, which have advanced maternal age (≥ 35) and seized for 14.4% of low prognosis, has a low cumulative live birth rate (11% in group 4). Female age is a critical element in the POSEIDON classification because age is crucially related to embryo ploidy and more importantly live birth outcome. The probability of having embryo ploidy sharply declined after the age of 34 and was lower than 50% in women aged 35 years and over. Therefore, patients in group 4 will have an increased risk of aneuploidy embryos, decreasing the live birth rate in these groups of patients. A recent study evaluated cumulative live birth rates per cycle, there was a remarkable difference between POSEIDON patients (21, 43, 10, 25, 29, and 17% in groups 1a, 1b, 2a, 2b, 3, and 4, respectively) and non-POSEIDON counterparts (52%). Facing difficulties related to clinical practice, optimizing the embryo culture process is necessary to improve the embryo number and quality in the POR group. Potential techniques include follicular size at the trigger, dual trigger, artificial oocyte activation (AOA), blastocyst transfer, and the role of preimplantation genetic testing for aneuploidy (PGT-A).

In Vietnam, AOA was first reported in 2011, performing on 1588 oocytes, and said the fertilization rate was higher in the ICSI - AOA than in the ICSI group (80.8% vs 74.3%, respectively; p<0.002).

AOA is expected to improve treatment outcomes for low prognosis patients, especially in group 4 by the POSEIDON criteria with the potential for clinical efficacy and safety. Therefore, this study aims to evaluate the effectiveness and safety of AOA on treatment outcomes in low prognosis patients defined by the POSEIDON criteria (2016).

ELIGIBILITY:
Inclusion Criteria:

* Was diagnosed as low prognosis patients by the POSEIDON criteria in group 4: maternal age ≥ 35 years old, AMH < 1,2 ng/ml and AFC < 5
* Cycles ≤ 3
* Oocytes could be collected with OPU procedure
* Ovarian stimulation with GnRH antagonist protocol
* Agree to participate in the randomization

Exclusion Criteria:

* Uterine abnormalities such as unicornuate, bicornuate uterus, didelphys and adenomyosis
* Recent history of any current untreated endocrine abnormality
* Gonadotropin resistance syndrome
* Contraindications of gonadotropins
* Absolute asthernozoospermia
* Cryptozoospermia
* Surgical sperm retrieval
* Previous low fertilization (< 30%)
* Globozoospermia
* Cycles using donor oocytes
* Preimplantation Genetic Testing (PGT) cycles

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women diagnosed as low prognosis patients by the POSEIDON criteria group 4 undergoing in vitro fertilization treatment.
Enrollment: 528 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | At 24 weeks of gestation
  The complete expulsion or extraction from a woman of a product of fertilisation, after 24 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 350 grams or more can be used if gestational age is unknown (twins are a single count).

SECONDARY OUTCOMES:
Fertilization rate | One day after oocyte retrieval
  The percentage of transformation of micro injected oocytes into two pronuclei
Fertilization failure rate | One day after oocyte retrieval
  The percentage transformation of micro injected oocytes into no pronuclei
Abnormal fertilization rate | One day after oocyte retrieval
  The percentage transformation of micro injected oocytes into more than two pronuclei
Total embryos on day 3 | Three days after oocyte retrieval
  Number of embryos on day 3
Good quality day 3 embryo rate | Three days after oocyte retrieval
  Number of good quality embryos on day 3
Total embryos blastocyst | Five days after oocyte retrieval
  Number of embryos on day 5
Good quality blastocyst rate | Five days after oocyte retrieval
  Number of good quality embryos on day 5
Positive pregnancy test | At 2 weeks after embryo placement
  Serum ß-hCG ≥25mIU/mL
Implantation rate | At 3 weeks after embryo placement
  Implantation rate is explained as as the number of gestational sacs per number of embryos transferred.
Cumulative implantation rate at 12 months | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative implantation rate.
  Cumulative implantation is total case of gestational sacs per total patient to be enrolled into the study at 12 months after randomization
Clinical pregnancy | At 7 weeks after embryo placement]
  Having at least 1 gestational sac on ultrasound at 5 weeks' gestation
Cumulative clinical pregnancy at 12 months | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative clinical pregnancy rate.
  Cumulative Clinical pregnancy is total case clinical pregnancy per total patient to be enrolled into the study at 12 months after randomization
Ongoing pregnancy | At 12 weeks after embryo placement
  Having at least 1 gestational sac on ultrasound at 12 weeks' gestation with heart beat activity
Cumulative ongoing pregnancy at 12 months | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative ongoing pregnancy rate.
  Cumulative ongoing pregnancy is total case ongoing pregnancy per total patient to be enrolled into the study at 12 months after randomization
Ectopic pregnancy | At 12 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualisation, or histopathology
Cumulative ectopic pregnancy at 12 months | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative ectopic pregnancy rate.
  Cumulative ectopic pregnancy is total case ectopic pregnancy per total patient to be enrolled into the study at 12 months after randomization
Miscarriage | At 12 weeks of gestation
  The spontaneous loss of an intra-uterine pregnancy prior to 12 completed weeks of gestational age
Cumulative miscarriage | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative miscarriage rate.
  Cumulative miscarriage is total case miscarriage per total patient to be enrolled into the study at 12 months after randomization
Multiple pregnancy | At 6 to 8 weeks' gestation
  ≥1 gestational sac at early pregnancy ultrasound
Cumulative multiple pregnancy | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative multiple pregnancy rate.
  Cumulative multiple pregnancy is total case multiple pregnancy per total patient to be enrolled into the study at 12 months after randomization
Vanishing twins | At 12 weeks' gestation
  Vanishing twins is defined as a pregnancy with two or more gestational sacs or positive heart beats at 7 weeks of gestation, but only one at 12 weeks' gestation.
Cumulative vanishing twins | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative vanishing twins rate.
  Cumulative vanishing twins is total case vanishing twins per total patient to be enrolled into the study at 12 months after randomization
Multiple delivery | At 24 weeks' gestation
  Birth of more than one baby beyond 24 weeks
Cumulative multiple delivery | 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative multiple delivery rate.
  Cumulative multiple delivery is total case multiple delivery per total patient to be enrolled into the study at 12 months after randomization
Hypertensive disorders of pregnancy | At 20 weeks of gestation or beyond after the completion of the first transfer
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Gestational diabetes mellitus | At 24 to 28 weeks of gestation
  using a 75g oral glucose tolerance test
Cumulative live birth rate | At 24 weeks of gestation
  Cumulative live birth rate at 12 months after the randomization.
Birth weight | At the time of delivery
  Weight of singletons and twins
Low birth weight | At birth
  Weight < 2500 gm at birth
Major congenital abnormalities | At birth
  Structural, functional, and genetic anomalies, that occur during pregnancy, and identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or are life-threatening, or cause death. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
High birth weight | At birth
  Weight >4000 gm at birth
Very low birth weight | At birth
  Weight < 1500 gm at birth
Large for gestational age | At birth
  defined as birth weight >90th centile for gestation, based on standardised ethnicity based charts
small for gestational age | At birth
  defined as less than 10th centile for gestational age at delivery based on standardised ethnicity based charts
Very high birth weight | At birth
  Weight >4500 gm at birth
Antepartum haemorrhage | At birth
  including placenta previa, placenta accreta and unexplained
Perinatal mortality | 24 weeks of gestation to the end of the neonatal period of 4 weeks after birth
  the death of a fetus or infant from 24 weeks of gestation to the end of the neonatal period of 4 weeks after birth.
Admission to NICU | At birth
  The admittance of the newborn to NICU

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, M.D, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- IVFMD, My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No